CLINICAL TRIAL: NCT06298071
Title: A Phase Ib Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Characteristics, and Initial Efficacy of Single and Multiple Dosing of Peguricase for Injection With Methotrexate in Patients With Gout.
Brief Title: A Phase Ib Clinical Trial of Peguricase for Injection With Methotrexate in Patients With Uncontrolled Gout.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIBP-R002-Ib
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Gout
Keywords: Uncontrolled gout; Peguricase for injection; Safety; Tolerability; Efficacy
MeSH Terms: conditions — Gout | interventions — Injections; Methotrexate

STUDY DESIGN:
Intervention Model Description: According to the sequence from low-dose group to high-dose group, there are 12 participants in each group, totaling 36 participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Injection; strength: 4mg.
  Interventions: Drug: SIBP-R002; Drug: Methotrexate
- Group 2 (Experimental): Injection; strength: 8mg.
  Interventions: Drug: SIBP-R002; Drug: Methotrexate
- Group 3 (Experimental): Injection; strength: 12mg.
  Interventions: Drug: SIBP-R002; Drug: Methotrexate

INTERVENTIONS:
Drug: SIBP-R002 — Injection; strength: 4mg. Each group consists of 12 participants. Firstly, 4 sentinel participants were enrolled in the single dose phase of peruricase for injection and methotrexate. After the sentinel participants completed a 5-day safety observation of the single dose, the remaining 8 participants in this group can be enrolled simultaneously. If there are no special circumstances, the participants in this group will enter the multi-dose stage of peruricase for injection combined with methotrexate within 2-4 weeks after completing a single dose.
  Other Names: Peguricase for injection
  Arms: Group 1
Drug: SIBP-R002 — Injection; strength: 8mg. Each group consists of 12 participants. Firstly, 4 sentinel participants were enrolled in the single dose phase of peruricase for injection and methotrexate. After the sentinel participants completed a 5-day safety observation of the single dose, the remaining 8 participants in this group can be enrolled simultaneously. If there are no special circumstances, the participants in this group will enter the multi-dose stage of peruricase for injection combined with methotrexate within 2-4 weeks after completing a single dose.
  Other Names: Peguricase for injection
  Arms: Group 2
Drug: SIBP-R002 — Injection; strength: 12mg. Each group consists of 12 participants. Firstly, 4 sentinel participants were enrolled in the single dose phase of peruricase for injection and methotrexate. After the sentinel participants completed a 5-day safety observation of the single dose, the remaining 8 participants in this group can be enrolled simultaneously. If there are no special circumstances, the participants in this group will enter the multi-dose stage of peruricase for injection combined with methotrexate within 2-4 weeks after completing a single dose.
  Other Names: Peguricase for injection
  Arms: Group 3
Drug: Methotrexate — Combination drugs: Methotrexate, dose15 mg, oral.

SUMMARY:
To evaluate the safety and tolerability of peguricase for injection with methotrexate in patients with gout who remain uncontrolled after standardized treatment with conventional uric acid-lowering drugs, to determine the recommended dose for phase II clinical trials, and to provide basis for formulation of administration regimen for phase II clinical trials.

DETAILED DESCRIPTION:
To evaluate the safety, tolerability, pharmacokinetics and pharmacodynamic characteristics, and initial efficacy of single and multiple dosing of peguricase for injection with methotrexate in patients with gout who remain uncontrolled after standardized treatment with conventional uric acid-lowering drugs.

This study is a phase Ib single and multiple dosing, dose-increasing. Three dose groups of 4, 8 or 12 mg were planned, then exploring the most appropriate dose for phase II clinical trials, and to provide basis for formulation of administration regimen for phase II clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent.
* Male and female aged between 18 and 70 years old , regardless of gender.
* Male weight ≥50 kg, female weight ≥45 kg, body mass index (BMI) in the range of (19-30) kg/m2 (including 19 and 30)；
* The clinical diagnosis of gout met the criteria of American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) in 2015，patients were in non-acute attack at screening or at least 2 weeks after complete remission of acute attack, and sUA ≥420 μmol/L at screening；
* Patients whose serum uric acid level could not reach the target after standard treatment with conventional uric acid-lowering drugs or who were contraindicated or intolerant to conventional uric acid-lowering drugs；
* Patients who were willing to stop taking any uric-acid-lowering drug at least 7 days before using methotrexate during the run-in period;
* Could tolerate the prescribed dose of methotrexate during the run-in period;
* Patients were able to attend and complete the visit on time.

Exclusion Criteria:

* Patients had active systemic infection within 2 weeks before enrollment，including an infection for which treatment was being received；
* Having a chronic or recurrent infection, such as recurrent pneumonia or chronic bronchitis; Patients with active or severe lung disease or pulmonary insufficiency on chest imaging, or current pulmonary fibrosis or bronchiectasis；
* Patients who are on anti-TB treatment or have active TB；
* Diagnosis of osteomyelitis；
* Ongoing or long-term use of immune system modulating drugs, such as methotrexate, mercaptopurine, mycophanolate, long-term use (≥3 months) of prednisone ≥10 mg/ day or equivalent dose of corticosteroids; Or have a history of transplant surgery requiring long-term immunotherapy; Or a known history of autoimmune disease, allergic disease;
* Known allergy to recombinant proteins or porcine products, or history of allergy to uricase, pegylated products, corticosteroids and antihistamines, or known intolerance to methotrexate, fexofenadine, acetaminophen or contraindications to methotrexate, fexofenadine, acetaminophen;
* Patients who are known to be intolerant to all gout attack management regiments (participants must be able to tolerate at least one: Colchicine and/or Nsaids and/or Prednisone 0.5 mg/kg daily；
* Patients who have previously been treated with pegyluricase or other recombinant uricase, or who have been treated with other pegylated biological products;
* Participation in other clinical study with a drug intervention within 4 weeks before initiation of methotrexate or the drug was still in the elimination phase before screening (within 5 half-lives), whichever is older;
* Patients with chronic liver disease such as hepatitis, cirrhosis, alcoholic liver disease;
* Patients have unstable angina, severe arrhythmias requiring drug intervention, congestive heart failure (NYHA grade≥Ⅱ), uncontrolled hypertension (over 150/95 mmHg), poor glycemic control in diabetics ( HbA1c≥7%), acute stroke, Severe or chronic hemorrhagic digestive disease, pleural and abdominal effusion;
* A history of hypoxanthine-guanine phosphoribosyltransferase deficiency, such as Lesch-Nyhan and Kelley-Seegmiller syndrome;
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency or G6PD test values below the lower limit of normal;
* Estimated glomerular filtration rate (eGFR) ≤40 mL/min/1.73m2, or currently receiving dialysis, or end-stage renal disease (CKD4-5);
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) above the upper limit of normal value or albumin below the lower limit of normal value during screening (before methotrexate treatment);
* Use of any blood component, short-acting or long-acting growth factor drugs within 14 days prior to screening, or white blood cell count < 4×109/L, hematopoietic volume < 32%, or platelet count < 75×109/L;
* Receiving anticoagulant therapy or international normalized ratio (INR) > 1.5×ULN or activated partial thromboplastin time (APTT) > 1.5×ULN before enrollment;
* Receiving systemic or local radiotherapy for tumors, or history of malignancy within 5 years other than non-melanoma skin cancer or in situ carcinoma of cervix;
* Any acute illness that was considered by the investigator to be likely to affect the study occurred within 1 month before screening;
* Donated (or lost) blood and donated (or lost) ≥400 mL or received blood transfusion within 3 months before screening;
* If any one of the five serological tests of hepatitis B was positive except for hepatitis B surface antibody, or hepatitis C antibody positive, treponema pallidum antibody positive or HIV antibody positive in serum virology examination;
* History of drug or substance abuse, or a positive drug screening test;
* History of alcohol abuse in the 3 months before screening [drinking more than 14 units of alcohol per week (1 unit ≈360 mL of beer)] or 45 mL of 40% spirits or 150 mL of wine)]; or positive alcohol breath test on admission;
* Lactating women, as well as male participants (or their partners) or female participants 30 days before the study to the end of the study, who have plans for pregnancy or sperm or egg donation within 6 months and are unwilling to take effective contraceptive measures;
* Patients have serious mental and psychological disorders, cognitive disorders and the existence of a history of mental illness.
* The investigator considered it inappropriate to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
AE(Adverse Events) | 14 weeks after the first dose
  That is adverse events, any adverse events that occurred to the participant during the study period.
SAE(Serious Adverse Events) | 14 weeks after the first dose
  That is serious adverse events, any serious adverse events that occurred to the participant during the study period.
AUC(Area Under The Plasma Concentration Versus Time Curve) | 14 weeks after the first dose
  It shows the degree to which a drug is absorbed and used in the body
Cmax(Peak Plasma Concentration) | 14 weeks after the first dose
  It shows the highest plasma concentration of a drug that can be achieved after administration.
Tmax(Peak Time) | 14 weeks after the first dose
  That is peak time of drug action, it shows the time required to reach the maximum concentration on the participant plasma concentration curve after administration.
T ½ (Terminal elimination half-life) | 14 weeks after the first dose
  It reflects how quickly the drug is eliminated from the body.
CL (Clearance Rate) | 14 weeks after the first dose
  Apparent volume of drug distribution removed from the body per unit time.
ADA (Anti-uricase Antibody, Anti-PEG Antibody, Anti-PEG-uricase Antibody) | 14 weeks after the first dose
  The incidence of anti-drug antibody.
NAb (Anti-PEG-uricase Neutralizing Antibody) | 14 weeks after the first dose
  The incidence of neutralizing antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhou, Master, Principal Investigator — Co., Ltd Shanghai Institute Of Biological Products
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No